CLINICAL TRIAL: NCT01664637
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Evaluation of the Efficacy and Safety of TZP-102 Given Orally Three Times a Day for the Treatment of Symptoms Associated With Diabetic Gastroparesis
Brief Title: Diabetic Gastroparesis Efficacy/Safety Study of TZP-102
Acronym: DIGEST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient efficacy in planned interim futility analysis
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TZP-102-CL-G004
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Diabetic Gastroparesis
Keywords: diabetic gastroparesis; delayed gastric emptying; gastroparesis; diabetes mellitus, Type 1; diabetes mellitus, Type 2
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TZP-102 three times a day (Experimental): 10 mg TZP-102 will be taken 30 minutes prior to each main meal for a total of three daily doses.
  Interventions: Drug: 10 mg TZP-102
- Placebo three times a day (Placebo Comparator): Placebo will be taken 30 minutes prior to each main meal for a total of three daily doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 10 mg TZP-102 — One oval-shaped, opaque-white, hard gelatin capsule containing active ingredient will be taken orally three times a day for 12 weeks
  Arms: TZP-102 three times a day
Drug: Placebo — One oval-shaped, opaque-white, hard gelatin capsule of placebo indistinguishable from active drug will be taken orally three times a day for 12 weeks
  Arms: Placebo three times a day

SUMMARY:
The purpose of this study is to test the safety and effectiveness of 10 mg TZP-102 given prior to meals three times a day compared to placebo (capsule that looks like active study drug but contains no active drug), administered for 12 weeks, in diabetic subjects with symptoms associated with gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age inclusive
* Type 1 or type 2 diabetes mellitus
* History of symptoms of gastroparesis for at least 3 months leading up to the Screening Visit
* Documented delayed gastric emptying
* Upper gastrointestinal obstruction ruled out by endoscopy or barium scan
* Concomitant medications must be stable for at least 2 weeks leading up to the Screening visit and must be maintained during the study.
* Females of child-bearing potential must have a negative serum pregnancy test and use (and agree to continue to use throughout the study) an acceptable form of contraception

Exclusion Criteria:

* Gastrectomy, bariatric surgery, fundoplication or vagotomy/pyloroplasty
* Has had or plans to have endoscopic pyloric injections of botulinum toxin within 6 months prior to the Screening Visit or during the study
* NG, PEG or PEJ feeding tube or inpatient hospitalization for gastroparesis within 2 weeks prior to the Screening Visit
* Required parenteral nutrition for treatment of gastroparesis within 2 months prior to the Screening Visit
* Active gastric pacemaker within 3 months prior to the Screening Visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symptoms associated with diabetic gastroparesis | 12 Weeks

SECONDARY OUTCOMES:
Change from baseline in health-related quality of life | 12 Weeks
Adverse events (AEs), vital signs, ECGs, clinical laboratory parameters | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Mondou, M.D., Study Director — Tranzyme, Inc.
Locations (32):
- United States (22):
  - Tranzyme Investigational Site, Huntsville, Alabama
  - Tranzyme Investigational Site, Tucson, Arizona
  - Tranzyme Investigational Site, North Little Rock, Arkansas
  - Tranzyme Investigational Site, Long Beach, California
  - Tranzyme Investigational Site, Ventura, California
  - Tranzyme Investigational Site, Hialeah, Florida
  - Tranzyme Investigational Site, Inverness, Florida
  - Tranzyme Investigational Site, Jacksonville, Florida
  - Tranzyme Investigational Site, Miami, Florida
  - Tranzyme Investigational Site, New Smyrna Beach, Florida
  - Tranzyme Investigational Site, Anderson, Indiana
  - Tranzyme Investigational Site, Indianapolis, Indiana
  - Tranzyme Investigational Site, Kansas City, Kansas
  - Tranzyme Investigational Site, Monroe, Louisiana
  - Tranzyme Investigational Site, Boston, Massachusetts
  - Tranzyme Investigational Site, Mexico, Missouri
  - Tranzyme Investigational Site, Raleigh, North Carolina
  - Tranzyme Investigational Site, Salisbury, North Carolina
  - Tranzyme Investigational Site, Winston-Salem, North Carolina
  - Tranzyme Investigational Site, Oklahoma City, Oklahoma
  - Tranzyme Investigational Site, Portland, Oregon
  - Tranzyme Investigational Site, El Paso, Texas
- Poland (10):
  - Tranzyme Investigational Site, Bialystok
  - Tranzyme Investigational Site, Bydgoszcz
  - Tranzyme Investigational Site, Kielce
  - Tranzyme Investigational Site, Krakow
  - Tranzyme Investigational Site, Lodz
  - Tranzyme Investigational Site, Lublin
  - Tranzyme Investigational Site, Olsztyn
  - Tranzyme Investigational Site, Rzeszów
  - Tranzyme Investigational Site, Warsaw
  - Tranzyme Investigational Site, Zgierz

REFERENCES:
- [Derived] McCallum RW, Lembo A, Esfandyari T, Bhandari BR, Ejskjaer N, Cosentino C, Helton N, Mondou E, Quinn J, Rousseau F; TZP-102 Phase 2b Study Group. Phase 2b, randomized, double-blind 12-week studies of TZP-102, a ghrelin receptor agonist for diabetic gastroparesis. Neurogastroenterol Motil. 2013 Nov;25(11):e705-17. doi: 10.1111/nmo.12184. Epub 2013 Jul 15. PMID 23848826